CLINICAL TRIAL: NCT02377362
Title: A 3-Part, Randomized, Double-Blind, Placebo-Controlled, Single and Multiple Ascending Dose, and Proof of Concept Study to Assess the Safety, Tolerability, Pharmacokinetics, and Pharmacodynamics of GLWL-01
Brief Title: A Study to Assess the Safety, Tolerability, Pharmacokinetics, and Pharmacodynamics of GLWL-01
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Insufficient efficacy for this indication. The study stopped after Part B.
Sponsor: GLWL Research Inc. (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: GLWL-SMP
Record Dates: First submitted 2015-02-25; First posted 2015-03-03 (Estimated); Results first posted 2019-03-21 (Actual); Last update posted 2019-03-21 (Actual); Status verified 2019-03

CONDITIONS: Diabetes Mellitus, Type 2
MeSH Terms: conditions — Diabetes Mellitus, Type 2

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (6):
- GLWL-01, Part A (Experimental): Escalating dose in at least 2 of 3 periods, starting at 10 milligrams (mg)
  Interventions: Drug: GLWL-01, Part A
- Placebo, Part A (Placebo Comparator): Escalating dose of placebo to match GLWL-01, in 1 period
  Interventions: Drug: Placebo, Part A
- GLWL-01, Part B (Experimental): Multiple ascending daily doses of GLWL-01 at up to six dose levels, based on Part A
  Interventions: Drug: GLWL-01, Part B
- Placebo, Part B (Placebo Comparator): Multiple daily doses of placebo to match GLWL-01
  Interventions: Drug: Placebo, Part B
- GLWL-01, Part C (Experimental): Multiple daily doses of GLWL-01 at level based upon Part B
  Interventions: Drug: GLWL-01, Part C
- Placebo, Part C (Placebo Comparator): Multiple daily doses of placebo to match GLWL-01
  Interventions: Drug: Placebo, Part C

INTERVENTIONS:
Drug: GLWL-01, Part A — Capsules administered orally, in 2 out of 3 periods
  Arms: GLWL-01, Part A
Drug: Placebo, Part A — Capsules administered orally in 1 out of 3 periods
  Arms: Placebo, Part A
Drug: GLWL-01, Part B — Capsules administered orally either once or twice daily for 27 days, with a single dose on Day 28
  Arms: GLWL-01, Part B
Drug: Placebo, Part B — Capsules administered orally either once or twice daily for 27 days with a single dose on Day 28
  Arms: Placebo, Part B
Drug: GLWL-01, Part C — Capsules administered orally either once or twice daily for 27 days with a single dose on Day 28
  Arms: GLWL-01, Part C
Drug: Placebo, Part C — Capsules administered orally either once or twice daily for 27 days with a single dose on Day 28
  Arms: Placebo, Part C

SUMMARY:
This 3-part study will explore the safety and tolerability of GLWL-01 in overweight/obese healthy participants after single doses (in Part A), and in participants with type 2 diabetes mellitus after multiple doses during a 28-day period (Parts B and C).

ELIGIBILITY:
Inclusion Criteria:

PARTS A-C:

* Non-vasectomized males (or those vasectomized less than 4 months prior to study start) must agree to use a condom with spermicide or abstain from sexual intercourse during the study until 90 days beyond the last dose of study drug
* Males agree to not donate sperm from dosing until 90 days after dosing
* Laboratory test results within normal range or acceptable deviation, and Aspartate Aminotransferase (AST) / Alanine Aminotransferase (ALT) / Gamma Glutamyl Transferase (GGT) / Alkaline Phosphatase (ALP) to be less than or equal to (≤)1.5 x upper limit of normal (ULN), and total bilirubin has to be within normal limit
* Estimated glomerular filtration rate (eGFR) greater than or equal to (≥) 60 milliliter (mL)/minute/1.73m2
* No evidence of weight excursion beyond 5% of baseline weight within 3 months of screening

PART A Only:

* Overtly healthy males or females, as determined by medical history and physical examination
* Males must be 18 to 65 years old; females must be 40 to 65 years old
* Female participants must be:

  1. Women with prior history of hysterectomy who are at least 45 years of age and with follicle-stimulating hormone (FSH) greater than (>) 40 milli-international units per milliliter (mIU/mL), or
  2. Menopausal women with either: spontaneous amenorrhea for at least 12 months (not induced by a medical condition or medications); or spontaneous amenorrhea for 6 to 12 months and a FSH > 40 mIU/mL
* Body mass index (BMI) of 28 to 35 kilograms divided by height in meters squared (kg/m2)
* Normotensive (supine systolic blood pressure (BP) less than (<) 140 millimeter of mercury (mmHg) and diastolic BP <90 mmHg
* No evidence of weight excursion beyond 5% of baseline weight within 3 months of screening

PARTS B and C:

* Must have Type 2 Diabetes Mellitus
* Be 18 to 70 years old
* Have BMI of 28 to 42 kg/m2
* Female participants must be of non-childbearing potential, and must have undergone one of the following sterilization procedures at least 6 months prior to first dose: hysteroscopic sterilization, bilateral tubal ligation or bilateral salpingectomy, hysterectomy, or bilateral oophorectomy; or be postmenopausal with amenorrhea for at least 1 year prior to the first dose and with FSH serum levels consistent with postmenopausal status
* Normotensive (supine systolic BP) < 150 mmHg and diastolic BP <95 mmHg or well-controlled hypertension while on a stable hypertensive

Exclusion Criteria:

PARTS A-C:

* Currently enrolled in a clinical trial or any other medical research judged to be not compatible with the study, or have participated in the last 30 days prior to dosing in a clinical trial involving an investigational product or non-approved use of a drug with short half-life, or within 5 half-lives of an investigational product with a half-life longer than 6 days
* Abnormality in the 12-lead electrocardiogram (ECG) including corrected QT (QTc) interval with Bazett's correction >450 milliseconds (msec) for men and >470 msec for women, or an abnormality that, in the opinion of the Investigator, increases the risks associated with participating in the study
* Significant cardiovascular disease or other disorders
* Evidence of human immunodeficiency virus (HIV) infection, hepatitis B, hepatitis C, or other chronic liver or biliary disease
* Average weekly alcohol intake that exceeds 21 units per week (males) and 14 units per week (females), or is unwilling to stop use of Cytochrome P450 (CYP3A) inhibitors/inducers (St. John's Wort) or alcohol consumption for the study, or regular use of known drugs of abuse or positive finding on urinary drug screen, use of cigarettes or nicotine products within last 3 months, or blood donation or loss within 56 days prior to the study
* Neuropsychiatric disease or pharmacological therapy for such conditions within 1 year of dosing, or antidepressants or antipsychotics within 3 months of dosing, or surgery within last 60 days
* Eating disorder or weight loss medications within 4 months of dosing, or bariatric surgery
* Unsuitable for inclusion in the study in the opinion of the investigator or sponsor

PART A Only:

* History of hypertension (or on treatment with any antihypertensives)
* Endocrine illness such as diabetes, growth hormone insufficiency / acromegaly, adrenal gland or thyroid illness

PARTS B and C:

* Currently taking simvastatin > 10 mg per day, or atorvastatin > 20 mg per day, or lovastatin >20 mg per day, or history of statin-induced myopathy / rhabdomyolysis. Participants taking any dose of simvastatin will be excluded from some cohorts
* Allergic to the components of the Mixed Meal Tolerance Test

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 74 (Actual)
Dates: Start 2015-03; Primary Completion 2016-11-09 (Actual); Study Completion 2016-11-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Email choruspharma@lists.lilly.com, Study Director — GLWL Research Inc.
Locations (4):
- United States (4):
  - Celerion, Tempe, Arizona
  - Profil Institute for Clinical Research, Inc., Chula Vista, California
  - Clinical Pharmacology of Miami, Inc., Miami, Florida
  - Clinical Trials of Texas, Inc., San Antonio, Texas

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Part A was a 3-period crossover design. Part A participants were to receive 2 escalating single doses of study drug and one dose of placebo. Part B participants were randomized to multiple doses of study drug or placebo. The study was stopped after Part B.
Groups:
- GLWL-01, Part A (Placebo; 150 mg; 600 mg): Part A: Cohort 1(C1) Sequence 1 (Placebo, 150 mg, 600 mg)
  Placebo was taken orally first intervention, then 150 mg GLWL 01 was taken orally second intervention, then 600 mg GLWL 01 was taken orally third intervention.
- GLWL-01, Part A (10 mg; Placebo; 600 mg): Part A: Cohort 1(C1) Sequence 2 (10 mg, Placebo, 600 mg)
  10 mg GLWL 01 was taken orally first intervention, then Placebo was taken orally second intervention, then 600 mg GLWL 01 was taken orally third intervention.
- GLWL-01, Part A (10 mg; 150 mg; Placebo): Part A: Cohort 1(C1) Sequence 3 (10 mg, 150 mg, Placebo)
  10 mg GLWL 01 was taken orally first intervention, then 150 mg GLWL 01 was taken orally second intervention, then Placebo was taken orally third intervention.
- GLWL-01, Part A (Placebo; 300 mg; 1200 mg): Part A: Cohort 2(C2) Sequence 1 (Placebo, 300 mg, 1200 mg)
  Placebo was taken orally first intervention, then 300 mg GLWL 01 was taken orally second intervention, then 1200 mg GLWL 01 was taken orally third intervention
- GLWL-01, Part A (50 mg, Placebo; 1200 mg): Part A: Cohort 2(C2) Sequence 2 (50 mg, Placebo, 1200 mg)
  50 mg GLWL 01 was taken orally first intervention, then Placebo was taken orally second intervention, then 1200 mg GLWL 01 was taken orally third intervention
- GLWL-01, Part A ( 50 mg; 300 mg; Placebo): Part A: Cohort 2(C3) Sequence 3 (50 mg, 300 mg, Placebo)
  50 mg GLWL 01 was taken orally first intervention, then 300 mg GLWL 01 was taken orally second intervention, then Placebo was taken orally third intervention.
- GLWL-01, Part B (50 mg, Twice a Day); GLWL-01, Part B (150 mg Twice a Day); GLWL-01, Part B (300 mg Once a Day); GLWL-01, Part B (450 mg Once a Day); GLWL-01, Part B, (450 mg Twice a Day); GLWL-01, Part B (600 mg Twice a Day): Multiple oral doses
  Part B: Capsules administered orally either once or twice daily for 27 days with a single dose on Day 28
- Placebo, Part B: Multiple oral doses of placebo to match GLWL-01
  Placebo, Part B: Capsules administered orally either once or twice daily for 27 days with a single dose on Day 28
Period: Part A First Treatment
Arm/Group | GLWL-01, Part A (Placebo; 150 mg; 600 mg) | GLWL-01, Part A (10 mg; Placebo; 600 mg) | GLWL-01, Part A (10 mg; 150 mg; Placebo) | GLWL-01, Part A (Placebo; 300 mg; 1200 mg) | GLWL-01, Part A (50 mg, Placebo; 1200 mg) | GLWL-01, Part A ( 50 mg; 300 mg; Placebo) | GLWL-01, Part B (50 mg, Twice a Day) | GLWL-01, Part B (150 mg Twice a Day) | GLWL-01, Part B (300 mg Once a Day) | GLWL-01, Part B (450 mg Once a Day) | GLWL-01, Part B, (450 mg Twice a Day) | GLWL-01, Part B (600 mg Twice a Day) | Placebo, Part B
Started | 4 | 4 | 4 | 4 | 4 | 4 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Completed | 4 | 4 | 4 | 4 | 4 | 4 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Period: Part A Second Treatment
Arm/Group | GLWL-01, Part A (Placebo; 150 mg; 600 mg) | GLWL-01, Part A (10 mg; Placebo; 600 mg) | GLWL-01, Part A (10 mg; 150 mg; Placebo) | GLWL-01, Part A (Placebo; 300 mg; 1200 mg) | GLWL-01, Part A (50 mg, Placebo; 1200 mg) | GLWL-01, Part A ( 50 mg; 300 mg; Placebo) | GLWL-01, Part B (50 mg, Twice a Day) | GLWL-01, Part B (150 mg Twice a Day) | GLWL-01, Part B (300 mg Once a Day) | GLWL-01, Part B (450 mg Once a Day) | GLWL-01, Part B, (450 mg Twice a Day) | GLWL-01, Part B (600 mg Twice a Day) | Placebo, Part B
Started | 4 | 4 | 4 | 4 | 4 | 4 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Completed | 4 | 4 | 4 | 4 | 3 | 4 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not Completed | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Protocol Violation | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Period: Part A Third Treatment
Arm/Group | GLWL-01, Part A (Placebo; 150 mg; 600 mg) | GLWL-01, Part A (10 mg; Placebo; 600 mg) | GLWL-01, Part A (10 mg; 150 mg; Placebo) | GLWL-01, Part A (Placebo; 300 mg; 1200 mg) | GLWL-01, Part A (50 mg, Placebo; 1200 mg) | GLWL-01, Part A ( 50 mg; 300 mg; Placebo) | GLWL-01, Part B (50 mg, Twice a Day) | GLWL-01, Part B (150 mg Twice a Day) | GLWL-01, Part B (300 mg Once a Day) | GLWL-01, Part B (450 mg Once a Day) | GLWL-01, Part B, (450 mg Twice a Day) | GLWL-01, Part B (600 mg Twice a Day) | Placebo, Part B
Started | 4 | 4 | 4 | 4 | 3 | 4 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Completed | 4 | 4 | 4 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not Completed | 0 | 0 | 0 | 4 | 3 | 4 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Highest dose level 1200 not used | 0 | 0 | 0 | 4 | 3 | 4 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Period: Part B Overall
Arm/Group | GLWL-01, Part A (Placebo; 150 mg; 600 mg) | GLWL-01, Part A (10 mg; Placebo; 600 mg) | GLWL-01, Part A (10 mg; 150 mg; Placebo) | GLWL-01, Part A (Placebo; 300 mg; 1200 mg) | GLWL-01, Part A (50 mg, Placebo; 1200 mg) | GLWL-01, Part A ( 50 mg; 300 mg; Placebo) | GLWL-01, Part B (50 mg, Twice a Day) | GLWL-01, Part B (150 mg Twice a Day) | GLWL-01, Part B (300 mg Once a Day) | GLWL-01, Part B (450 mg Once a Day) | GLWL-01, Part B, (450 mg Twice a Day) | GLWL-01, Part B (600 mg Twice a Day) | Placebo, Part B
Started (Part A was a 3-period crossover study (2 escalating doses of GLWL and 1 dose of placebo)) | 0 | 0 | 0 | 0 | 0 | 0 | 6 | 6 | 6 | 7 | 6 | 7 | 12
Completed | 0 | 0 | 0 | 0 | 0 | 0 | 4 | 5 | 6 | 6 | 6 | 6 | 12
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 1 | 0 | 1 | 0 | 1 | 0
Not completed — Protocol Violation | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Not completed — Adverse Event | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0
Not completed — Withdrawal by Subject | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0

BASELINE CHARACTERISTICS:
Population: .Part A was a crossover design. Part A participants were to receive 2 escalating doses of study drug and one dose of placebo in 3 periods.
Groups:
- GLWL-01 Part A (50 mg, Placebo; 1200 mg): Part A: Cohort 2(C2) Sequence 2 (50 mg, Placebo, 1200 mg)
  50 mg GLWL 01 was taken orally first intervention, then Placebo was taken orally second intervention, then 1200 mg GLWL 01 was taken orally third intervention
- GLWL-01, Part B (50 mg Twice a Day); GLWL-01, Part B (150 mg Twice a Day); GLWL-01, Part B (300 mg Once a Day); GLWL-01, Part B (450 mg Once a Day); GLWL-01, Part B (450 mg Twice a Day); GLWL-01, Part B (600 mg Twice a Day): Multiple oral doses
  Part B: Capsules administered orally either once or twice daily for 27 days with a single dose on Day 28
- Total: Total of all reporting groups
Arm/Group | GLWL-01, Part A (Placebo; 150 mg; 600 mg) | GLWL-01, Part A (10 mg; Placebo; 600 mg) | GLWL-01, Part A (10 mg; 150 mg; Placebo) | GLWL-01, Part A (Placebo; 300 mg; 1200 mg) | GLWL-01 Part A (50 mg, Placebo; 1200 mg) | GLWL-01, Part A ( 50 mg; 300 mg; Placebo) | GLWL-01, Part B (50 mg Twice a Day) | GLWL-01, Part B (150 mg Twice a Day) | GLWL-01, Part B (300 mg Once a Day) | GLWL-01, Part B (450 mg Once a Day) | GLWL-01, Part B (450 mg Twice a Day) | GLWL-01, Part B (600 mg Twice a Day) | Placebo, Part B | Total
Number analyzed (Participants) | 4 | 4 | 4 | 4 | 4 | 4 | 6 | 6 | 6 | 7 | 6 | 7 | 12 | 74
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 4 | 4 | 4 | 4 | 4 | 4 | 6 | 5 | 6 | 5 | 4 | 6 | 10 | 66
  >=65 years | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 2 | 2 | 1 | 2 | 8
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 0 | 0 | 1 | 0 | 0 | 1 | 2 | 2 | 3 | 4 | 4 | 8 | 27
  Male | 2 | 4 | 4 | 3 | 4 | 4 | 5 | 4 | 4 | 4 | 2 | 3 | 4 | 47
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2 | 1 | 1 | 3 | 2 | 4 | 4 | 4 | 5 | 5 | 6 | 7 | 12 | 56
  Not Hispanic or Latino | 2 | 3 | 3 | 1 | 2 | 0 | 2 | 2 | 1 | 2 | 0 | 0 | 0 | 18
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2
  Asian | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 1 | 1 | 5
  White | 4 | 3 | 3 | 3 | 4 | 4 | 5 | 4 | 6 | 7 | 6 | 6 | 11 | 66
  More than one race | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 4 | 4 | 4 | 4 | 4 | 4 | 6 | 6 | 6 | 7 | 6 | 7 | 12 | 74

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With One or More Treatment Emergent Adverse Events (Part A)
Description: Treatment Emergent Adverse Event defined as an adverse event that started or worsened in severity at the time of, or after treatment
Time Frame: Baseline to 7 weeks
Measure: Count of Participants; unit: Participants
Groups:
- GLWL-01 Part A (10mg): 10 milligrams (mg)
- GLWL-01 Part A (50 mg): 50 mg
- GLWL-01 Part A (150 mg): 150 mg
- GLWL-01 Part A (300 mg): 300 mg
- GLWL-01 Part A (600 mg): 600 mg
Arm/Group | GLWL-01 Part A (10mg) | GLWL-01 Part A (50 mg) | GLWL-01 Part A (150 mg) | GLWL-01 Part A (300 mg) | GLWL-01 Part A (600 mg) | GLWL-01 Part A Placebo
Number analyzed (Participants) | 8 | 8 | 8 | 8 | 8 | 19
Participants | 1 | 2 | 0 | 2 | 3 | 9

2. Primary Outcome: Number of Participants With One or More Treatment Emergent Adverse Events (Parts B)
Description: as for outcome 1
Time Frame: Baseline to 6 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | GLWL-01 Part B (50 mg, Twice a Day) | GLWL-01 Part B (150 mg, Twice a Day) | GLWL-01 Part B (300 mg, Once a Day) | GLWL-01 Part B (450 mg, Once a Day) | GLWL-01 Part B (450 mg, Twice a Day) | GLWL-01 Part B (600 mg, Twice a Day) | GLWL-01 Part B Placebo
Number analyzed (Participants) | 6 | 6 | 6 | 7 | 6 | 7 | 12
Participants | 5 | 5 | 3 | 5 | 4 | 7 | 6

3. Secondary Outcome: Area Under the Plasma Concentration-Time Curve From Time Zero to the Last Non-Zero Concentration (AUC0-t) (Part A)
Time Frame: Pre-dose, 0.5, 1, 2, 4.5, 6, 8.5, 12.5, 24, 28.5, 48, 96 and 144 hours post-dose
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: µg*hr/mL
Arm/Group | GLWL-01 Part A (10mg) | GLWL-01 Part A (50 mg) | GLWL-01 Part A (150 mg) | GLWL-01 Part A (300 mg) | GLWL-01 Part A (600 mg)
Number analyzed (Participants) | 8 | 8 | 8 | 8 | 8
µg*hr/mL | 0.5119 (15.7) | 3.138 (13.7) | 12.91 (38.2) | 35.16 (16.9) | 118.8 (32.9)

4. Secondary Outcome: Area Under the Plasma Concentration-Time Curve From Time Zero to the Last Non-Zero Concentration (AUC0-t) (Part B)
Time Frame: Predose, 0.5, 1, 2, 4.5, 6, 8.5, 12, 13, 14, 16, 24, 48, 168, and 336 hours post dose starting on Day 28
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng*hr/mL
Groups:
- GLWL-01 Part B (50mg, Twice a Day): 50 milligrams (mg), twice a day (BID)
- GLWL-01 Part B (150 mg, Twice a Day): 150 mg, twice a day (BID)
- GLWL-01 Part B (300 mg, Once a Day): 300 mg, once a day (QD)
- GLWL-01 Part B (450 mg, Once a Day): 450 mg once a day (QD)
- GLWL-01 Part B (450 mg, Twice a Day): 450 mg twice a day (BID)
- GLWL-01 Part B (600 mg, Twice a Day): 600 mg, twice a day (BID)
Arm/Group | GLWL-01 Part B (50mg, Twice a Day) | GLWL-01 Part B (150 mg, Twice a Day) | GLWL-01 Part B (300 mg, Once a Day) | GLWL-01 Part B (450 mg, Once a Day) | GLWL-01 Part B (450 mg, Twice a Day) | GLWL-01 Part B (600 mg, Twice a Day)
Number analyzed (Participants) | 4 | 5 | 6 | 6 | 6 | 6
ng*hr/mL | 5040 (30.6) | 37000 (22.5) | 47500 (17.1) | 124000 (41.9) | 202000 (26.6) | 235000 (39.2)

5. Secondary Outcome: Area Under the Plasma Concentration-Time Curve From Time Zero to 24-hour Post-Dose (AUC0-24) (Part A)
Time Frame: Predose, 0.5, 1, 2, 4.5, 6, 8.5, 12, 13, 14, 16, 24 hours post-dose
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: µg*hr/mL
Arm/Group | GLWL-01 Part A (10mg) | GLWL-01 Part A (50 mg) | GLWL-01 Part A (150 mg) | GLWL-01 Part A (300 mg) | GLWL-01 Part A (600 mg)
Number analyzed (Participants) | 8 | 8 | 8 | 8 | 8
µg*hr/mL | 0.551 (16.5) | 3.15 (11.6) | 12.6 (38.0) | 34.4 (16.9) | 110 (29.4)

6. Secondary Outcome: Area Under the Plasma Concentration-Time Curve From Time Zero to 24-hour Post-Dose (AUC0-24) (Parts B)
Time Frame: Predose, 0.5, 1, 2, 4.5, 6, 8.5, 12, 13, 14, 16, 24 hours post dose starting on Day 28
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng*hr/mL
Arm/Group | GLWL-01 Part B (50mg, Twice a Day) | GLWL-01 Part B (150 mg, Twice a Day) | GLWL-01 Part B (300 mg, Once a Day) | GLWL-01 Part B (450 mg, Once a Day) | GLWL-01 Part B (450 mg, Twice a Day) | GLWL-01 Part B (600 mg, Twice a Day)
Number analyzed (Participants) | 4 | 5 | 6 | 6 | 6 | 6
ng*hr/mL | 5040 (30.6) | 34600 (21.7) | 45700 (16.9) | 111000 (39.0) | 184000 (25.2) | 210000 (37.7)

7. Secondary Outcome: Area Under the Plasma Concentration-Time Curve From Time Zero to Infinity (AUC0-inf) (Part A)
Time Frame: Pre-dose, 0.5, 1, 2, 4.5, 6, 8.5, 12.5, 24, 28.5, 48, 96 and 144 hours post-dose
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: µg*hr/mL
Arm/Group | GLWL-01 Part A (10mg) | GLWL-01 Part A (50 mg) | GLWL-01 Part A (150 mg) | GLWL-01 Part A (300 mg) | GLWL-01 Part A (600 mg)
Number analyzed (Participants) | 8 | 8 | 8 | 8 | 8
µg*hr/mL | 0.555 (16.7) | 3.19 (12.1) | 13.0 (41.2) | 35.4 (17.5) | 119 (32.7)

8. Secondary Outcome: Area Under the Plasma Concentration-Time Curve From Time Zero to Infinity (AUC0-inf) (Part B)
Time Frame: Predose, 0.5, 1, 2, 4.5, 6, 8.5, 12, 13, 14, 16, 24, 48, 168, and 336 hours post dose starting Day 1
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng*hr/mL
Arm/Group | GLWL-01 Part B (50mg, Twice a Day) | GLWL-01 Part B (150 mg, Twice a Day) | GLWL-01 Part B (300 mg, Once a Day) | GLWL-01 Part B (450 mg, Once a Day) | GLWL-01 Part B (450 mg, Twice a Day) | GLWL-01 Part B (600 mg, Twice a Day)
Number analyzed (Participants) | 6 | 6 | 6 | 7 | 6 | 7
ng*hr/mL | 3150 (20.1) | 13500 (14.8) | 31800 (21.9) | 69300 (31.4) | 79000 (19.5) | 127000 (16.0)

9. Secondary Outcome: Maximum Observed Drug Concentration (Cmax) (Part A)
Time Frame: Pre-dose, 0.5, 1, 2, 4.5, 6, 8.5, 12.5, 24, 28.5, 48, 96 and 144 hours post-dose
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: µg/mL
Arm/Group | GLWL-01 Part A (10mg) | GLWL-01 Part A (50 mg) | GLWL-01 Part A (150 mg) | GLWL-01 Part A (300 mg) | GLWL-01 Part A (600 mg)
Number analyzed (Participants) | 8 | 8 | 8 | 8 | 8
µg/mL | 0.121 (8.4) | 0.600 (35.4) | 2.47 (39.9) | 5.08 (17.6) | 11.5 (23.9)

10. Secondary Outcome: Maximum Observed Drug Concentration (Cmax) (Part B)
Time Frame: Predose, 0.5, 1, 2, 4.5, 6, 8.5, 12, 13, 14, 16, 24, 48, 168, and 336 hours post dose starting on Day 28
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | GLWL-01 Part B (50mg, Twice a Day) | GLWL-01 Part B (150 mg, Twice a Day) | GLWL-01 Part B (300 mg, Once a Day) | GLWL-01 Part B (450 mg, Once a Day) | GLWL-01 Part B (450 mg, Twice a Day) | GLWL-01 Part B (600 mg, Twice a Day)
Number analyzed (Participants) | 4 | 5 | 6 | 6 | 6 | 6
ng/mL | 785 (45.8) | 37.90 (28.1) | 62.80 (10.6) | 10800 (31.5) | 16300 (25.9) | 18200 (33.7)

11. Secondary Outcome: Time to Observed Cmax (Tmax) (Part A)
Time Frame: Pre-dose, 0.5, 1, 2, 4.5, 6, 8.5, 12.5, 24, 28.5, 48, 96 and 144 hours post-dose
Measure: Median (Full Range); unit: hours
Arm/Group | GLWL-01 Part A (10mg) | GLWL-01 Part A (50 mg) | GLWL-01 Part A (150 mg) | GLWL-01 Part A (300 mg) | GLWL-01 Part A (600 mg)
Number analyzed (Participants) | 8 | 8 | 8 | 8 | 8
hours | 1.00 [0.999 to 1.02] | 1.51 [0.476 to 4.50] | 1.02 [0.466 to 4.55] | 1.50 [1.00 to 4.50] | 1.00 [0.998 to 6.00]

12. Secondary Outcome: Time to Observed Cmax (Tmax) (Part B)
Time Frame: Predose, 0.5, 1, 2, 4.5, 6, 8.5, 12, 13, 14, 16, 24, 48, 168, and 336 hours post dose starting on Day 28
Measure: Median (Full Range); unit: hours
Arm/Group | GLWL-01 Part B (50mg, Twice a Day) | GLWL-01 Part B (150 mg, Twice a Day) | GLWL-01 Part B (300 mg, Once a Day) | GLWL-01 Part B (450 mg, Once a Day) | GLWL-01 Part B (450 mg, Twice a Day) | GLWL-01 Part B (600 mg, Twice a Day)
Number analyzed (Participants) | 4 | 5 | 6 | 6 | 6 | 6
hours | 2.00 [1.00 to 4.5] | 2.00 [2.00 to 4.5] | 1.00 [0.99 to 2.00] | 3.25 [0.999 to 6.00] | 2.00 [1.00 to 4.50] | 4.5 [2.00 to 4.5]

13. Secondary Outcome: Elimination Half-Life (T1/2) (Part A)
Time Frame: Pre-dose, 0.5, 1, 2, 4.5, 6, 8.5, 12.5, 24, 28.5, 48, 96 and 144 hours post-dose
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: hours
Arm/Group | GLWL-01 Part A (10mg) | GLWL-01 Part A (50 mg) | GLWL-01 Part A (150 mg) | GLWL-01 Part A (300 mg) | GLWL-01 Part A (600 mg)
Number analyzed (Participants) | 8 | 8 | 8 | 8 | 8
hours | 3.32 (8.8) | 3.77 (23.9) | 5.22 (25.3) | 5.25 (25.8) | 5.47 (19.0)

14. Secondary Outcome: Elimination Half-Life (T1/2) (Part B)
Time Frame: Predose, 0.5, 1, 2, 4.5, 6, 8.5, 12, 13, 14, 16, 24, 48, 168, and 336 hours post dose starting on Day 28
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: hours
Arm/Group | GLWL-01 Part B (50mg, Twice a Day) | GLWL-01 Part B (150 mg, Twice a Day) | GLWL-01 Part B (300 mg, Once a Day) | GLWL-01 Part B (450 mg, Once a Day) | GLWL-01 Part B (450 mg, Twice a Day) | GLWL-01 Part B (600 mg, Twice a Day)
Number analyzed (Participants) | 4 | 5 | 6 | 6 | 6 | 6
hours | 5.33 (12.1) | 6.16 (15.16) | 5.24 (20.3) | 5.94 (14.9) | 5.12 (18.5) | 6.26 (16.7)

15. Secondary Outcome: Apparent Clearance of Drug (CL/F) (Part A)
Time Frame: Pre-dose, 0.5, 1, 2, 4.5, 6, 8.5, 12.5, 24, 28.5, 48, 96 and 144 hours post-dose
Measure: Mean (Standard Deviation); unit: L/hr
Arm/Group | GLWL-01 Part A (10mg) | GLWL-01 Part A (50 mg) | GLWL-01 Part A (150 mg) | GLWL-01 Part A (300 mg) | GLWL-01 Part A (600 mg)
Number analyzed (Participants) | 8 | 8 | 8 | 8 | 8
L/hr | 18.27 (3.17) | 15.78 (2.18) | 12.16 (4.16) | 8.59 (1.37) | 5.27 (1.77)

16. Secondary Outcome: Apparent Clearance of Drug (CL/F) (Part B)
Time Frame: Predose, 0.5, 1, 2, 4.5, 6, 8.5, 12, 13, 14, 16, 24, 48, 168, and 336 hours post dose starting on Day 28
Measure: Mean (Standard Deviation); unit: L/hr
Arm/Group | GLWL-01 Part B (50mg, Twice a Day) | GLWL-01 Part B (150 mg, Twice a Day) | GLWL-01 Part B (300 mg, Once a Day) | GLWL-01 Part B (450 mg, Once a Day) | GLWL-01 Part B (450 mg, Twice a Day) | GLWL-01 Part B (600 mg, Twice a Day)
Number analyzed (Participants) | 4 | 5 | 6 | 6 | 6 | 6
L/hr | 11.4 (3.57) | 5.20 (1.14) | 6.64 (1.10) | 4.27 (1.35) | 3.23 (0.76) | 3.97 (1.36)

17. Secondary Outcome: Apparent Total Volume of Distribution (VZ/F) (Part A)
Time Frame: Pre-dose, 0.5, 1, 2, 4.5, 6, 8.5, 12.5, 24, 28.5, 48, 96 and 144 hours post-dose
Measure: Mean (Standard Deviation); unit: L
Arm/Group | GLWL-01 Part A (10mg) | GLWL-01 Part A (50 mg) | GLWL-01 Part A (150 mg) | GLWL-01 Part A (300 mg) | GLWL-01 Part A (600 mg)
Number analyzed (Participants) | 8 | 8 | 8 | 8 | 8
L | 86.87 (10.765) | 86.35 (15.326) | 88.09 (17.282) | 66.97 (20.368) | 41.43 (13.114)

18. Secondary Outcome: Apparent Total Volume of Distribution (VZ/F) (Part B)
Time Frame: Predose, 0.5, 1, 2, 4.5, 6, 8.5, 12, 13, 14, 16, 24, 48, 168, and 336 hours post dose starting on Day 28
Measure: Mean (Standard Deviation); unit: L
Arm/Group | GLWL-01 Part B (50mg, Twice a Day) | GLWL-01 Part B (150 mg, Twice a Day) | GLWL-01 Part B (300 mg, Once a Day) | GLWL-01 Part B (450 mg, Once a Day) | GLWL-01 Part B (450 mg, Twice a Day) | GLWL-01 Part B (600 mg, Twice a Day)
Number analyzed (Participants) | 4 | 5 | 6 | 6 | 6 | 6
L | 89.6 (39.15) | 46.3 (10.18) | 51.2 (14.76) | 36.8 (12.39) | 24.2 (7.055) | 35.8 (12.01)

19. Secondary Outcome: Amount of Drug Excreted in Urine (Aet1-t12) (Part A)
Description: Data Not Collected for this Parameter
Time Frame: Pre-Dose and 12 hours Post-Dose
Population: Data were not collected
Arm/Group | GLWL-01 Part A (10mg) | GLWL-01 Part A (50 mg) | GLWL-01 Part A (150 mg) | GLWL-01 Part A (300 mg) | GLWL-01 Part A (600 mg) | GLWL-01 Part A Placebo
Number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0

20. Secondary Outcome: Amount of Drug Excreted in Urine (Aet1-t12) (Part B)
Description: Data Not Collected for this Parameter
Time Frame: Pre-Dose and 12 hours Post-Dose on Day 28
Population: Data were not collected
Arm/Group | GLWL-01 Part B (50 mg, Twice a Day) | GLWL-01 Part B (150 mg, Twice a Day) | GLWL-01 Part B (300 mg, Once a Day) | GLWL-01 Part B (450 mg, Once a Day) | GLWL-01 Part B (450 mg, Twice a Day) | GLWL-01 Part B (600 mg, Twice a Day) | GLWL-01 Part B Placebo
Number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0

21. Secondary Outcome: Amount of Drug Excreted in Urine (Aet0-24) (Part A)
Time Frame: Pre-Dose and 24-hours Post-Dose
Measure: Mean (Standard Deviation); unit: mg
Arm/Group | GLWL-01 Part A (10mg) | GLWL-01 Part A (50 mg) | GLWL-01 Part A (150 mg) | GLWL-01 Part A (300 mg) | GLWL-01 Part A (600 mg)
Number analyzed (Participants) | 7 | 8 | 8 | 8 | 8
mg | 1.87 (0.611) | 11.7 (2.56) | 36.9 (12.1) | 101 (15.2) | 191 (37.4)

22. Secondary Outcome: Amount of Drug Excreted in Urine (Aet0-24) (Part B)
Time Frame: Pre-Dose and 24-hours Post-Dose on Day 28
Measure: Mean (Standard Deviation); unit: mg
Arm/Group | GLWL-01 Part B (50mg, Twice a Day) | GLWL-01 Part B (150 mg, Twice a Day) | GLWL-01 Part B (300 mg, Once a Day) | GLWL-01 Part B (450 mg, Once a Day) | GLWL-01 Part B (450 mg, Twice a Day) | GLWL-01 Part B (600 mg, Twice a Day)
Number analyzed (Participants) | 4 | 5 | 6 | 6 | 6 | 6
mg | 28.2 (12.87) | 94.8 (9.843) | 125 (33.45) | 175 (25.93) | 272 (67.08) | 293 (77.33)

23. Secondary Outcome: Fraction of Drug Excreted in the Urine (Fe) (Part A)
Time Frame: Pre-Dose and 24-hours Post-Dose
Measure: Mean (Standard Deviation); unit: percentage of the drug
Arm/Group | GLWL-01 Part A (10mg) | GLWL-01 Part A (50 mg) | GLWL-01 Part A (150 mg) | GLWL-01 Part A (300 mg) | GLWL-01 Part A (600 mg)
Number analyzed (Participants) | 7 | 8 | 8 | 8 | 8
percentage of the drug | 18.7 (6.11) | 23.3 (5.13) | 24.6 (8.08) | 33.6 (5.07) | 31.8 (6.23)

24. Secondary Outcome: Fraction of Drug Excreted in the Urine (Fe) (Part B)
Time Frame: Pre-Dose and 24-hours Post-Dose on Day 28
Measure: Mean (Standard Deviation); unit: percentage of the drug
Arm/Group | GLWL-01 Part B (50mg, Twice a Day) | GLWL-01 Part B (150 mg, Twice a Day) | GLWL-01 Part B (300 mg, Once a Day) | GLWL-01 Part B (450 mg, Once a Day) | GLWL-01 Part B (450 mg, Twice a Day) | GLWL-01 Part B (600 mg, Twice a Day)
Number analyzed (Participants) | 4 | 5 | 6 | 6 | 6 | 6
percentage of the drug | 56.3 (25.74) | 63.2 (6.562) | 41.5 (11.15) | 38.9 (5.761) | 60.5 (14.91) | 48.9 (12.89)

25. Secondary Outcome: Change From Baseline in Average Plasma Glucose Concentration After Multiple Doses (Part B)
Time Frame: Baseline to Day 24-26
Population: The 450 mg twice a day arm had no usable continuous glucose data, due to technical difficulties
Measure: Mean (Standard Deviation); unit: mg/dL
Groups:
- GLWL-01, Part B (450 mg Twice a Day): 450 mg twice a day (BID)
Arm/Group | GLWL-01 Part B (50mg, Twice a Day) | GLWL-01 Part B (150 mg, Twice a Day) | GLWL-01 Part B (300 mg, Once a Day) | GLWL-01 Part B (450 mg, Once a Day) | GLWL-01, Part B (450 mg Twice a Day) | GLWL-01 Part B (600 mg, Twice a Day) | Placebo Part B
Number analyzed (Participants) | 5 | 4 | 6 | 4 | 0 | 6 | 9
mg/dL | 22.53 (23.0) | 7.38 (40.4) | 7.92 (30.3) | 21.39 (13.5) |  | 5.43 (38.0) | 8.05 (41.9)

26. Secondary Outcome: Change From Baseline in Postprandial Glucose (Part B)
Description: Mixed Meal Tolerance Test (4.5 hours after a meal on Day 28); Baseline Adjusted. The day 28 values were used for analysis; change from baseline was calculated on Day 28.
Time Frame: Day 28
Measure: Mean (Standard Deviation); unit: mg/dL
Groups:
- GLWL-01, Part B (450 mg, Twice a Day): 450 mg, twice a day (BID)
Arm/Group | GLWL-01 Part B (50mg, Twice a Day) | GLWL-01 Part B (150 mg, Twice a Day) | GLWL-01 Part B (300 mg, Once a Day) | GLWL-01 Part B (450 mg, Once a Day) | GLWL-01, Part B (450 mg, Twice a Day) | GLWL-01 Part B (600 mg, Twice a Day) | Placebo Part B
Number analyzed (Participants) | 4 | 5 | 6 | 6 | 6 | 6 | 12
mg/dL | 18.8 (11.70) | 11.6 (27.74) | -13.7 (33.16) | 10.7 (27.40) | 29.3 (49.43) | 29.7 (25.77) | 13.2 (41.41)

27. Secondary Outcome: Change From Baseline in C-Peptide Concentration (Part B)
Description: Mixed Meal Tolerance Test (4.5 hours after a meal on Day 28); Baseline-Adjusted. The day 28 values were used for analysis; change from baseline was calculated on Day 28.
Time Frame: Day 28
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | GLWL-01 Part B (50mg, Twice a Day) | GLWL-01 Part B (150 mg, Twice a Day) | GLWL-01 Part B (300 mg, Once a Day) | GLWL-01 Part B (450 mg, Once a Day) | GLWL-01, Part B (450 mg, Twice a Day) | GLWL-01 Part B (600 mg, Twice a Day) | Placebo Part B
Number analyzed (Participants) | 3 | 5 | 6 | 6 | 6 | 6 | 11
ng/mL | 0.373 (0.257) | 0.338 (0.9523) | 0.437 (0.5171) | 0.575 (1.0658) | 0.360 (1.3600) | 0.457 (0.8498) | 0.043 (0.6513)

28. Secondary Outcome: Change From Baseline in Insulin Concentration (Part B)
Description: 4.5 hours following Mixed Meal Tolerance Test (MMTT) on Day 28; Baseline Adjusted. The day 28 values were used for analysis; change from baseline was calculated on Day 28.
Time Frame: Day 28
Measure: Mean (Standard Deviation); unit: uU/mL
Groups:
- GLWL-01 Part B (450 mg, Twice a Day): 450 mg, twice a day (BID)
Arm/Group | GLWL-01 Part B (50mg, Twice a Day) | GLWL-01 Part B (150 mg, Twice a Day) | GLWL-01 Part B (300 mg, Once a Day) | GLWL-01 Part B (450 mg, Once a Day) | GLWL-01 Part B (450 mg, Twice a Day) | GLWL-01 Part B (600 mg, Twice a Day) | Placebo Part B
Number analyzed (Participants) | 3 | 5 | 6 | 6 | 6 | 6 | 11
uU/mL | -3.60 (7.579) | -3.89 (11.533) | -9.75 (10.687) | 2.12 (5.878) | 1.27 (9.194) | 0.23 (7.653) | 2.39 (8.263)

29. Secondary Outcome: Fasting Glucose Concentration (Part B)
Description: Fasting glucose concentration after 28 day treatment
Time Frame: Baseline to Day 28
Measure: Mean (Standard Deviation); unit: mmol/L
Arm/Group | GLWL-01 Part B (50mg, Twice a Day) | GLWL-01 Part B (150 mg, Twice a Day) | GLWL-01 Part B (300 mg, Once a Day) | GLWL-01 Part B (450 mg, Once a Day) | GLWL-01 Part B (450 mg, Twice a Day) | GLWL-01 Part B (600 mg, Twice a Day) | Placebo Part B
Number analyzed (Participants) | 4 | 5 | 3 | 4 | 6 | 6 | 10
mmol/L | 1.15 (1.139) | 1.10 (1.520) | -0.20 (2.100) | 0.63 (0.299) | -1.13 (1.381) | -0.10 (2.104) | 0.91 (2.116)

30. Secondary Outcome: Change From Baseline in Weight (Part B)
Time Frame: Baseline to Day 28
Measure: Mean (Standard Deviation); unit: kilograms (kg)
Arm/Group | GLWL-01 Part B (50mg, Twice a Day) | GLWL-01 Part B (150 mg, Twice a Day) | GLWL-01 Part B (300 mg, Once a Day) | GLWL-01 Part B (450 mg, Once a Day) | GLWL-01 Part B (450 mg, Twice a Day) | GLWL-01 Part B (600 mg, Twice a Day) | Placebo Part B
Number analyzed (Participants) | 4 | 5 | 6 | 6 | 6 | 6 | 12
kilograms (kg) | -0.375 (0.763) | -0.340 (0.786) | -0.150 (0.995) | -0.417 (0.741) | 0.417 (1.229) | 0.350 (0.356) | -0.025 (0.717)

31. Secondary Outcome: Change From Baseline in Waist Circumference (Part B)
Time Frame: Baseline to Day 28
Measure: Mean (Standard Deviation); unit: centimeters
Arm/Group | GLWL-01 Part B (50mg, Twice a Day) | GLWL-01 Part B (150 mg, Twice a Day) | GLWL-01 Part B (300 mg, Once a Day) | GLWL-01 Part B (450 mg, Once a Day) | GLWL-01 Part B (450 mg, Twice a Day) | GLWL-01 Part B (600 mg, Twice a Day) | Placebo Part B
Number analyzed (Participants) | 4 | 5 | 6 | 6 | 6 | 6 | 12
centimeters | -1.275 (3.522) | 1.360 (5.755) | -3.517 (4.001) | -1.383 (5.123) | -1.250 (1.091) | -0.083 (0.492) | -0.867 (4.026)

32. Secondary Outcome: Change From Baseline in Hip Circumference (Part B)
Time Frame: Baseline to Day 28
Measure: Mean (Standard Deviation); unit: centimeters
Arm/Group | GLWL-01 Part B (50mg, Twice a Day) | GLWL-01 Part B (150 mg, Twice a Day) | GLWL-01 Part B (300 mg, Once a Day) | GLWL-01 Part B (450 mg, Once a Day) | GLWL-01 Part B (450 mg, Twice a Day) | GLWL-01 Part B (600 mg, Twice a Day) | Placebo Part B
Number analyzed (Participants) | 4 | 5 | 6 | 6 | 6 | 6 | 12
centimeters | -1.05 (2.940) | 0.960 (7.442) | 1.283 (2.337) | -0.417 (2.094) | 0.167 (0.753) | -0.333 (0.516) | 0.192 (6.860)

ADVERSE EVENTS:
Groups:
- GLWL-01, Part A (10mg): 10 milligrams (mg)
Arm/Group | GLWL-01, Part A (10mg) | GLWL-01 Part A (50 mg) | GLWL-01 Part A (150 mg) | GLWL-01 Part A (300 mg) | GLWL-01 Part A (600 mg) | GLWL-01 Part A Placebo | GLWL-01 Part B (50 mg, Twice a Day) | GLWL-01 Part B (150 mg, Twice a Day) | GLWL-01 Part B (300 mg, Once a Day) | GLWL-01 Part B (450 mg, Once a Day) | GLWL-01 Part B (450 mg, Twice a Day) | GLWL-01 Part B (600 mg, Twice a Day) | GLWL-01 Part B Placebo
All-Cause Mortality (participants affected / at risk) | 0/8 | 0/8 | 0/8 | 0/8 | 0/8 | 0/19 | 0/6 | 0/6 | 0/6 | 0/7 | 0/6 | 0/7 | 0/12
Serious Adverse Events (participants affected / at risk) | 0/8 | 0/8 | 0/8 | 0/8 | 0/8 | 0/19 | 0/6 | 0/6 | 0/6 | 0/7 | 0/6 | 0/7 | 0/12
Other Adverse Events (participants affected / at risk) | 1/8 | 2/8 | 0/8 | 2/8 | 3/8 | 9/19 | 5/6 | 5/6 | 3/6 | 5/7 | 4/6 | 7/7 | 6/12
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | GLWL-01, Part A (10mg) (N=8) | GLWL-01 Part A (50 mg) (N=8) | GLWL-01 Part A (150 mg) (N=8) | GLWL-01 Part A (300 mg) (N=8) | GLWL-01 Part A (600 mg) (N=8) | GLWL-01 Part A Placebo (N=19) | GLWL-01 Part B (50 mg, Twice a Day) (N=6) | GLWL-01 Part B (150 mg, Twice a Day) (N=6) | GLWL-01 Part B (300 mg, Once a Day) (N=6) | GLWL-01 Part B (450 mg, Once a Day) (N=7) | GLWL-01 Part B (450 mg, Twice a Day) (N=6) | GLWL-01 Part B (600 mg, Twice a Day) (N=7) | GLWL-01 Part B Placebo (N=12)
Diarrhoea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 2 (4) | 1 (6) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 4 (4)
Nausea (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 2 (2) | 2 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 1 (2)
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Abdominal pain lower (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dyspepsia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Eructation (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 1 (1)
Flatulence (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0)
Headache (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 3 (3) | 2 (5) | 0 (0) | 1 (1) | 2 (3) | 0 (0) | 4 (4) | 1 (1)
Dizziness postural (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 2 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Paraesthesia (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Catheter site pain (General disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Catheter site paraesthesia (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Skin abrasion (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Decreased appetite (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 4 (4) | 1 (1)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pallor (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Vision blurred (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Visual impairment (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Viral upper respiratory tract infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Vomiting (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Abdominal Discomfort (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Abdominal Distension (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Faeces Discolored (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Faeces Soft (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Haematochezia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Toothache (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dizziness (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Hypoglycaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Myalgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (3) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Back Pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Limb Discomfort (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Musculoskeletal Discomfort (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Musculoskeletal Pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pain in Extremity (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Fatigue (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Vessel Puncture Site Pain (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Medical Device Site Haemorrhage (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Oedema Peripheral Pain (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Vessel Puncture Site Haemorrhage (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Vessel Puncture Site Induration (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Urinary Tract Infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Otitis Media (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Upper Respiratory Tract Infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Nasopharyngitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Blood Glucose Increase (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (3) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Blood Creatine Phosphokinase Increase (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Aspartate Aminotransferase Increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Blood Lactate Dehydrogenase Increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Eye Irritation (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pollakiuria (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Tachycardia (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Palpitations (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Anxiety (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Rhinitis Allergic (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Palmar Erythema (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pain (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Rhinitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes